CLINICAL TRIAL: NCT01234298
Title: A Phase 3 Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Low- and High-dose Range Groups of SPD489 as Adjunctive Treatment to Established Maintenance Doses of Antipsychotic Medications on Negative Symptoms in Clinically Stable Adults Who Have Persistent Predominant Negative Symptoms of Schizophrenia
Brief Title: SPD489 as Adjunctive Treatment in Adults With Negative Symptoms of Schizophrenia
Acronym: NSS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was discontinued due to non-safety related business prioritization decisions
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD489-320
Record Dates: First submitted 2010-10-29; First posted 2010-11-04 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Negative Symptoms of Schizophrenia
MeSH Terms: interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- SPD489 Low-Dose (Experimental)
  Interventions: Drug: SPD489 Low-Dose
- SPD489 High-Dose (Experimental)
  Interventions: Drug: SPD489 High-Dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPD489 Low-Dose — SPD489 20, 30, or 40 mg capsules taken once-daily for up to 26 weeks
  Other Names: Vyvanse, Lisdexamfetamine dimesylate, LDX
  Arms: SPD489 Low-Dose
Drug: SPD489 High-Dose — SPD489 50, 60, or 70 mg capsules taken once-daily for up to 26 weeks
  Other Names: Vyvanse, Lisdexamfetamine dimesylate, LDX
  Arms: SPD489 High-Dose
Drug: Placebo — Placebo capsule taken once-daily for up to 26 weeks
  Arms: Placebo

SUMMARY:
To assess the safety and efficacy of SPD489 low-dose and high-dose treatment groups to placebo when given as adjunctive therapy to antipsychotic medication in clinically stable adults with persistent predominant negative symptoms of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Subject has diagnosis of schizophrenia for at least 2 years
* Subject has persistent predominant negative symptoms
* Subject has 2 or more persistent predominant negative symptoms (affective flattening, alogia, avolition apathy, and anhedonia-asociality) determined to have been present for at least 6 months
* Subject is maintained on antipsychotic monotherapy or polytherapy with no more than 2 antipsychotic medications
* Subject has been clinically stable and is in the non-acute phase of illness

Exclusion Criteria:

* Subject has clinically notable positive symptoms
* Subject is considered to be treatment refractory
* Subject has current history of substance abuse/dependance
* Subject is considered a suicide risk or risk to harm others

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01-27 (Estimated); Primary Completion 2014-02-24 (Estimated); Study Completion 2014-02-24 (Estimated)

PRIMARY OUTCOMES:
Negative Symptom Assessment (NSA-16) total score | up to 26 weeks

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | up to 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda